CLINICAL TRIAL: NCT05659121
Title: Evaluating Evidence-based and Sustainable Application of Robotic Exoskeletons in Rehabilitation for Those With Impaired Mobility
Brief Title: Improving Mobility Via Robotic Exoskeletons in Local Rehabilitation Settings in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Temasek Foundation Cares (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iMOVE
Record Dates: First submitted 2022-04-14; First posted 2022-12-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Spinal Cord Injuries; Spinal Cord Diseases
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EksoGT group (Experimental): Participants in the intervention group will receive 12 sessions of robotic exoskeleton training incorporated into their conventional physiotherapy session.
  Interventions: Device: robotic exoskeleton training
- Control group (No Intervention): Participants in the control group will only undergo outcome measures assessment. They will continue with their conventional physiotherapy and the frequency and type of activity at physiotherapy will be recorded.

INTERVENTIONS:
Device: robotic exoskeleton training — robotic exoskeleton training using EksoGT will be incorporated into subject's conventional physiotherapy training.
  Arms: EksoGT group

SUMMARY:
The programme is designed to investigate the application of robotic exoskeleton in different levels of local rehabilitation facilities. Feasibilities, efficacy, cost-effectiveness, patient and therapist's view of the application of robotic exoskeleton will be evaluated.

DETAILED DESCRIPTION:
In recent years, robot-assisted gait training has been increasingly applied in various rehabilitation facilities across Singapore. Thus far, all systems in Singapore are tethered to treadmills or other platforms. These are bulky, expensive, and the 'gait' trained differs from normal gait to varying degrees. Such systems are found only in hospitals and major centres with significant space and financial resources. No evaluation of cost-effectiveness has been performed thus far. With appropriate and efficient clinical protocols adapted and optimised for the Singapore context, study team plans to demonstrate engaging and cost-effective delivery of rehabilitation care, particularly in the community. The aims of the programme include:

1. To study the feasibility of the robotic exoskeleton application in both hospital and community rehabilitation settings (inpatient and outpatient)
2. To investigate if robotic exoskeletons training could improve motor outcomes in patients with impaired mobility, in the subacute and chronic phases of recovery.
3. To evaluate the cost-effectiveness of robotic exoskeleton application in rehabilitation.

400 participants with impaired walking ability will be recruited at a 3:1 ratio (intervention: control) from participating centres of the iMOVE programme (Improving Mobility Via Exoskeletons) in Singapore. The iMOVE Programme is a pilot clinical programme, funded by Temasek Foundation Cares, evaluating the utility of robotic exoskeletons for the rehabilitation of mobility across the continuum of rehabilitation care.

This will be a non-randomized controlled study. Eligible participants will be asked for their willingness to undergo robotic exoskeleton training (RET). Those who decline intervention will be offered participation in the control group, where they will receive their usual care with conventional physiotherapy.

Participants in the intervention group will receive 12 sessions of RET incorporated into their conventional physiotherapy session. Typical total duration of physiotherapy is 45-60 minutes, comprising 30 minutes of RET, and 15-30 minutes of conventional physiotherapy. The training period will follow participant's own physiotherapy schedule, the frequency of which might range from 5 times a week (for inpatient) to 1-2 times a week (for outpatient). Outcome measures including measurement for functional mobility and quality of life will be performed before training, after training and 6 months post-training.

Participants in the control group will only undergo outcome measures assessment. They will continue with their conventional physiotherapy and the frequency and type of activity at physiotherapy will be recorded. Outcome measures for the control group will be performed at similar time points as the intervention group, i.e., before training (i.e., after signing ICF), after training (after 12 sessions of conventional physiotherapy) and 6 months later.

The application of robotic exoskeleton in rehabilitation among patients with walking impairment will also be evaluated through qualitatively exploring the perceptions of patients and therapists. The factors influencing the utilization of the robotic exoskeletons for rehabilitation among patients will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 to 90 years old;
2. Functional Ambulatory Category (FAC) 0-3;
3. Able to follow instructions adequately to ensure safe use of the exoskeleton.

Exclusion Criteria

1. Severe osteoporosis;
2. Uncontrolled medical conditions (eg. Unstable angina, untreated hypertension);
3. Terminal disease with expected survival <1 year;
4. Pressure sores or wounds at point of contact with exoskeleton;
5. Severe limitations of range of movement in the lower limb (eg. from contractures or spasticity);
6. Lower limb fractures that have not been fixed or are deemed not stable enough for training with exoskeleton;
7. Cognitive impairment so as to be unable to follow instructions;
8. Significant pain in the lower limbs.
9. Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Functional ambulatory category | baseline
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Higher score indicates better ambulation ability.
Functional ambulatory category | up to 12 weeks
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Higher score indicates better ambulation ability.
Functional ambulatory category | 6 months
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Higher score indicates better ambulation ability.
10 meter walk test | baseline
  Test for walking speed
10 meter walk test | up to 12 weeks
  Test for walking speed
10 meter walk test | 6 months
  Test for walking speed
6 minute walk test | baseline
  Test for walking endurance. Distance covered in 6 minutes with participant's comfortable walking speed will be recorded.
6 minute walk test | up to 12 weeks
  Test for walking endurance. Distance covered in 6 minutes with participant's comfortable walking speed will be recorded.
6 minute walk test | 6 months
  Test for walking endurance. Distance covered in 6 minutes with participant's comfortable walking speed will be recorded.
Walking Index for Spinal Cord Injury | baseline
  It is tested for patient with spinal cord injury only. It assess the amount of physical assistance needed, as well as device required, for walking following paralysis that results from Spinal Cord Injury. Scale ranges from 0 to 20. Higher scores mean a better outcome, i.e. less assistance required.
Walking Index for Spinal Cord Injury | up to 12 weeks
  It is tested for patient with spinal cord injury only. It assess the amount of physical assistance needed, as well as device required, for walking following paralysis that results from Spinal Cord Injury. Scale ranges from 0 to 20. Higher scores mean a better outcome, i.e. less assistance required.
Walking Index for Spinal Cord Injury | 6 months
  It is tested for patient with spinal cord injury only. It assess the amount of physical assistance needed, as well as device required, for walking following paralysis that results from Spinal Cord Injury. Scale ranges from 0 to 20. Higher scores mean a better outcome, i.e. less assistance required.
clinical outcome variables scale (COVS) (for non-walkers) | baseline
  The COVS is an assessment scale used to quantify functional mobility status. It contains 13 items. Each item is scored on a 7-point scale ranging from 1 (fully dependent mobility) to 7 (normal independent mobility). Higher scores mean a higher mobility function.
clinical outcome variables scale (COVS) (for non-walkers) | up to 12 weeks
  The COVS is an assessment scale used to quantify functional mobility status. It contains 13 items. Each item is scored on a 7-point scale ranging from 1 (fully dependent mobility) to 7 (normal independent mobility). Higher scores mean a higher mobility function.
clinical outcome variables scale (COVS) (for non-walkers) | 6 months
  The COVS is an assessment scale used to quantify functional mobility status. It contains 13 items. Each item is scored on a 7-point scale ranging from 1 (fully dependent mobility) to 7 (normal independent mobility). Higher scores mean a higher mobility function.
Cycle ergometer testing | baseline
  This test is for non-walkers.
Cycle ergometer testing | up to 12 weeks
  This test is for non-walkers.
Cycle ergometer testing | 6 months
  This test is for non-walkers.
Goal Attainment Scale | baseline
  The Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met. Each patient effectively has their own outcome measures, but these measures are scored in a standardized way: +2: much more than expected; +1: somewhat more than expected; 0: patient achieves the expected level; -1: somewhat less than expected; -2: much less than expected. The overall score is calculated by incorporating the goal scores into a single aggregated t-score.
Goal Attainment Scale | up to 12 weeks
  TThe Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met. Each patient effectively has their own outcome measures, but these measures are scored in a standardized way: +2: much more than expected; +1: somewhat more than expected; 0: patient achieves the expected level; -1: somewhat less than expected; -2: much less than expected. The overall score is calculated by incorporating the goal scores into a single aggregated t-score.
Goal Attainment Scale | 6 months
  The Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met. Each patient effectively has their own outcome measures, but these measures are scored in a standardized way: +2: much more than expected; +1: somewhat more than expected; 0: patient achieves the expected level; -1: somewhat less than expected; -2: much less than expected. The overall score is calculated by incorporating the goal scores into a single aggregated t-score. selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met.

SECONDARY OUTCOMES:
Rivermead mobility index | baseline
  Assess functional mobility in gait, balance and transfers after stroke. It consists of 15 items. The items are scored 0 if the patient is not able to complete the task or 1 if they are able to complete it. The points are then added together, to score a maximum of 15, with higher scores stipulating better functional mobility.
Rivermead mobility index | up to 12 weeks
  Assess functional mobility in gait, balance and transfers after stroke. It consists of 15 items. The items are scored 0 if the patient is not able to complete the task or 1 if they are able to complete it. The points are then added together, to score a maximum of 15, with higher scores stipulating better functional mobility.
Rivermead mobility index | 6 months
  Assess functional mobility in gait, balance and transfers after stroke. It consists of 15 items. The items are scored 0 if the patient is not able to complete the task or 1 if they are able to complete it. The points are then added together, to score a maximum of 15, with higher scores stipulating better functional mobility.
EuroQol-5 dimension (EQ5D) | baseline
  EQ-5D is a standardised measure of health-related quality of life. It consists of 5 dimensions of health- mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimensions scores from 1 to 5, with 1 indicating "no problems" and 5 indicating "being unable to do' or extreme pain/discomfort/anxiety/depression.
EuroQol-5 dimension (EQ5D) | 6 months
  EQ-5D is a standardised measure of health-related quality of life. It consists of 5 dimensions of health- mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimensions scores from 1 to 5, with 1 indicating "no problems" and 5 indicating "being unable to do' or extreme pain/discomfort/anxiety/depression.
7-day physical activity recall | baseline
  for outpatient only
7-day physical activity recall | up to 12 weeks
  for outpatient only
7-day physical activity recall | 6 months
  for outpatient only
RET satisfaction survey and feedback | up to 12 weeks
  For the intervention group only. Each question is scaled from 1 to 7, with 1 indicating the most negative response, while 7 indicating the most positive response.
Technology Awareness Survey | baseline
  It contains 15 questions designed by the study team, to explore participants' initial view on the application of innovative technology such as robotic exoskeleton in rehabilitation, before they start the physiotherapy with RET. The result is not reported in ordinal scale.

OTHER OUTCOMES:
semi-structured interview | up to 12 weeks
  To explore the perceptions of the robotic exoskeleton and the factors influencing the utilization of robotic exoskeletons for rehabilitation among users.

CONTACTS AND LOCATIONS:
Overall Officials: Effie Chew, MBBS, Principal Investigator — Senior Consultant
Locations (2):
- Singapore (2):
  - Alexandra Hospital, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shankar R, Tang N, Shafawati N, Phan P, Mukhopadhyay A, Chew E. Cost-effectiveness analysis of robotic exoskeleton versus conventional physiotherapy for stroke rehabilitation in Singapore from a health system perspective. BMJ Open. 2025 Jul 7;15(7):e095269. doi: 10.1136/bmjopen-2024-095269. PMID 40623888
- [Derived] Tam PK, Tang N, Kamsani NSB, Yap TY, Coffey-Aladdin I, Goh SM, Tan JPP, Lui YC, Lee RL, Suresh R, Chew E. Overground robotic exoskeleton vs conventional therapy in inpatient stroke rehabilitation: results from a pragmatic, multicentre implementation programme. J Neuroeng Rehabil. 2025 Jan 6;22(1):3. doi: 10.1186/s12984-024-01536-1. PMID 39762953